Cover page with the Official Title of the study:

Effectiveness of the Transdiagnostic Treatment in the Population of Tijuana and Juarez with

Anxiety and Electrophysiological Correlation Measurements. A Randomized Clinical Trial.

Date: November 15th of 2018

Informed Consent Form (ICF)



## **INFORMED CONSENT LETTER**

PROGRAM: EFFECTIVENESS OF THE TRANSDIAGNOSTIC TREATMENT IN THE POPULATION OF TIJUANA AND JUAREZ WITH ANXIETY AND ELECTROPHYSIOLOGICAL CORRELATION MEASUREMENTS. A RANDOMIZED CLINICAL TRIAL

| NAME OF THE PARTICIPANT: |
|-----------------------------------|
| DATE OF SIGNINF INFORMED CONSENT: |
| NUMBER OF THE REGISTER: |

**Purpose:** The objective of the research is to validate the efficacy of a psychological treatment based on scientific evidence for the treatment of a wide range of anxiety disorders. As well as observing the modification of activity in the frontal symmetry before and after the treatment.

**Procedure:** The study includes the application of various instruments oriented towards the detection of anxious symptoms such as:

- EMOTIVE EPOC + of 14 channels.
- Post-Traumatic Stress Disorder (PTSD) Symptom Scale (PSS) (Foa, Riggs, Dancu y Rothbaum, 1993).
- Interview Program for Anxiety Disorders. (Brown, DiNardo y Barlow, 1994).
- Beck Depression Inventory. (Beck, Steer y Brown, 1996).
- State Trait Anxiety Inventory (1975, 2007).
- Generalized Anxiety Disorder 7-item (GAD-7) scale (Spitzet, 2006).
- Big Five Inventory (Oliver, 2008).
- Scale of Beck's Suicidal Ideation. (Beck, Kovacs y Weissman, 1979).
- Scale of therapeutic alliance negotiation (Peña Leyva, 2016).

You will receive a treatment based on the transdiagnostic model, which includes the implementation of 8 modules distributed from 11 to 17 sessions, with a duration of one hour each.

Risks and Discomforts: No risk or discomfort has been detected in the participation in this research.

Confidentiality: The data of the participants will be treated with confidentiality, and destroyed once the study has concluded and after 5 years.

Benefits: Receive psychological treatment based on scientific evidence, without cost.

Participation: Your participation in this program is voluntary and can be withdrawn at any time you wish. If you wish to withdraw from the program, please notify the researcher in advance.

If you have any doubt, question or disagreement, you can clarify it with the person in charge of the project, Dr. Alejandro Domínguez Rodríguez, at his mail, alejandro.dominguez.rodriguez@uabc.edu.mx or Dr. Graciela Avitia at her email graciela.avitia@uacj.mx

| Name and signature of the participant | Name and signature of whom obtains the consent |
|---|---|

Witness 1 Witness 2

Name, address, relationship and signature

Name, address, relationship and signature